#### NCT03259360

#### UNIVERSITY OF CALIFORNIA, SAN FRANCISCO CONSENT TO BE IN RESEARCH

**Study Title:** The Put it Out Project (POP)

| Research Project | Danielle Ramo, Ph.D., Assistant Professor in Residence. |
|---|---|
| Director: | UCSF, Phone: |
| Study Coordinator: | Lauren Smith, M.S., Clinical Research Coordinator Phone: |

The Put it Out Project (POP) is a clinical research study and it is voluntary.

Research studies include only people who choose to take part. Please take your time to make your decision about participating. You may discuss your decision with your family and friends or with your health care team. If you have any questions, you may ask the study staff.

You are being asked to take part in this study because you are a young adult who identifies as lesbian, gay, bisexual, transgender, or questioning (LGBTQ+) and smokes cigarettes.

The lead researcher, Danielle Ramo Ph.D., from the University of California, San Francisco and study staff are available to explain the study to you or to answer questions. They can be reached at \_\_or

## Why Is This Study Being done?

This study is helping researchers to evaluate two social media interventions for tobacco use with LGBTQ+ young adults.

# How many people are participating in this study?

At least 120 people will participate in this study.

#### Am I eligible to participate in the study?

To participate in the POP study, you need to be between 18 and 25 years old today, identify as sexual or gender minority (i.e., LGBTQ+), and smoke cigarettes.

#### What will happen if I take part in this study?

If you agree to participate in this study you will be asked to complete three surveys and join a secret Facebook group, where you will be asked to comment on 90 posts over 90 days and participate in weekly live sessions with a counselor.

If you agree to participate and provide contact information you will be sent the first survey. The survey asks about some of the things you may have done recently, like smoking or drinking, how you use social media, demographic information (e.g., age, ethnic background, school and employment history, illegal drug use), and some thoughts or experiences you've had about sexuality and homophobia. It will take you about 20 minutes to complete the survey.

Once you have completed the survey, you will be "randomized" into one of the study groups described below. Randomization means that you are put into a group by chance. A computer program will place you in one of the groups. Neither you nor the study staff can choose the group you will be in. You will have an equal chance of being placed in either group. If you are interested and eligible, you will be invited to a completely private ("secret") Facebook group where we will conduct the group with participants like yourself and our study staff. You will be asked to remain in the group for 90 days and comment on one of our posts once a day for three whole months.

Study participants will be assigned at random to one of the two study groups, described below:

### If you are in Group 1...

Participants in the Group 1 will be invited to a private group on Facebook along with other people who feel the same way about smoking as they do. We will let you know when the group will officially begin. POP staff will make daily posts to the group for 90 days and you are encouraged to join in the discussions, but your participation is completely voluntary. There will also be times when you can talk directly with a tobacco cessation counselor through the secret groups if you choose. You will have access to the secret group for 6 months from the day you join the group.

#### If you are in Group 2...

Participants in Group 2 will be invited to a different type of private Facebook group along with other people who feel the same way about smoking as they do. We will let you know when the group will officially begin. POP staff will make daily posts to the group for 90 days that are tailored to LGBTQ+ populations and you are encouraged to join in the discussions, but your participation is completely voluntary. The posts will be different than in Group 1. There will also be times when you can talk directly with a tobacco cessation counselor through the secret groups if you choose. You will have access to the secret group for 6 months from the day you join the group.

After the active part of the group is over (90 days) we will ask you to complete a survey. This survey will ask you some questions about what you liked or disliked about being in the Facebook group, and some other questions about your smoking. If, upon completing this survey, you report that you have quit smoking we will ask you for you postal address in order to send you a saliva test kit to confirm that you have indeed quit

smoking. We will ask you to complete the test kit and email or Facebook message us a picture of the test results.

Another three months after that we will ask you to complete a similar survey for your final task as a participant in our study (about 6 months from now.) If, upon completing this survey, you report that you have quit smoking we will ask you to complete another saliva test kit and send us your results via email or Facebook messenger.

## How long?

You will be enrolled in the study for 6 months; our study asks you to remain in a private Facebook group for three months, where we will ask you to respond to one post a day, estimating that you may spend about 5-10 minutes a day for 90 days. You will also be asked to complete 3 surveys, one at the start of the program, one end of program survey, and another survey 3 months after that. Each of the three surveys will take about 20-30 minutes to complete.

## Are there any risks to me or my privacy?

Participation in research can cause a loss of privacy. The researchers will keep information about you as confidential as possible, but due to the nature of Facebook, complete confidentiality cannot be guaranteed. Additionally, University of California may look at Research Records after the study is complete.

Although we will do our best to protect your study information (see below), there is still a risk of loss of privacy. Any information that you disclose on Facebook as part of this study may be shown to others in your Facebook network, depending on your privacy settings and the terms of agreement dictated by Facebook. Furthermore, although Facebook groups are entirely private, participation in the group may make your Facebook profile name known to other users who are also part of the study. Your Facebook profile name will not be connected to your survey responses in any way. The completed surveys will be kept secure and separate from information which identifies you including your name, email, and phone number. Only a small number of researchers will have direct access to completed surveys. If this study is published or presented at scientific meetings, names and other information that might identify you will not be used.

Each person can only complete each survey one time. In order to help us make sure this happens, we will also keep track of your computer's IP address. The IP address will not be linked to your survey data in any way.

In order to send you the surveys to complete, and to send you compensation for study participation, we will ask for your email address and phone number if you agree to participate in the study. If you give us your email address and/or phone number, we may send you a secure, encrypted email or text message asking you to complete each survey. The email address or phone number you provide will not be linked to your survey data.

There may be some discomfort associated with change in tobacco use if you decide to do so during the course of this study.

Finally, some of the survey and/or group questions may make you feel uncomfortable or raise unpleasant memories. You are free to stop the surveys or the group at any time.

### **Certificate of Confidentiality**

To help us protect your privacy, we have obtained a Certificate of Confidentiality from the National Institutes of Health. With this Certificate, the researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings.

Exceptions: A Certificate of Confidentiality does not prevent researchers from voluntarily disclosing information about you, without your consent. For example, we will voluntarily disclose information about incidents such as child abuse, and intent to hurt yourself or others. In addition, a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. If an insurer, employer, or other person obtains your written consent to receive research information, then the researchers may not use the Certificate to withhold that information. Finally, the Certificate may not be used to withhold information from the Federal government needed for auditing or evaluating federally funded projects or information needed by the FDA.

### Are there benefits to taking part in the study?

You may benefit by changing your smoking habits, and perhaps eventually quitting smoking, but this cannot be guaranteed. However, the information that you provide may help health professionals better understand/learn more about tobacco use with LGBTQ+ young adults through social networking sites.

#### Can I say "No"?

Yes, you do not have to complete any surveys or participate in the secret groups. If you choose not to be in this study you will not lose any of your regular benefits, and you can still receive medical care from UCSF if you are a patient.

#### Are there any payments or costs?

There are no costs for participating in this study.

## Will I be paid for taking part in the study?

You are able to earn a total of \$170 in Amazon gift cards sent via email for participating in this study. You may receive \$20 for completing the initial survey, \$90 for commenting on all of the 90 posts on Facebook over 90 days, \$20 for completing the survey at the end of the 90 days, and finally another \$20 for completing our final survey after another three months. If you complete all three surveys you will earn a bonus \$20 for a total of \$80.

What are my rights if I take part in the study?



Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you in any way. You will not lose any of your regular benefits, and you can still get your care from our institution the way you usually do.

## Who can answer my questions about the study?



If you wish to ask questions about the study or your rights as a research participant to someone other than the researchers or if you wish to voice any problems or concerns you may have about the study, please call the Institutional Review Board at 415-476-1814 or email at irb@ucsf.edu.

Thank you for considering our study. Your participation is greatly appreciated.

Please check one of the boxes below:

- o Yes, I agree to participate in this survey.
- No thanks, I would not like to participate.